CLINICAL TRIAL: NCT05824793
Title: The Efficacy of A-PRF+ on Postoperative Outcomes Following Surgical Removal of Impacted Mandibular Third Molars: a Randomized Controlled Trial
Brief Title: The Efficacy of A-PRF+ on Postoperative Outcomes Following Surgical Removal of Impacted Mandibular Third Molars (A-PRF+: Advanced Platelet Rich Fibrin)
Acronym: A-PRF+
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Nguyen Thi Bich Ly, Senior Lecturer/Dr, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 194/ĐHYD-HĐĐĐ
Record Dates: First submitted 2023-03-25; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: PRF
Keywords: Impacted mandibular third molar; tooth extraction; A-PRF+; pain; trismus; swelling
MeSH Terms: conditions — Pain; Trismus

STUDY DESIGN:
Intervention Model Description: Each patient enrolled in the research was encoded using a code from 001 to n, in blocks of 10 numbers, compared to the number on the sealed envelope with the random number pre-selected via the function RAND() on Microsoft Excel by the data collector. Number in the patient's envelope: odd number of group 1, even number of group 2. In case the patient has two IMTM that need to be extracted, meeting the inclusion and exclusion criteria of the study; after random: if the first time in the odd group, be operated on according to the standard procedure, the remaining opposite teeth would be surgically operated on using A-PRF+, the second time after the first surgery at least five weeks. And similarly, if randomly selecting the number is an even.
  * Control group (group 1 = odd number): no use of A-PRF+ after tooth extraction.
  * Study group (group 2 = even number): use A-PRF+ after tooth extraction.
Who Masked: Outcomes Assessor
Masking Description: Each participant was assigned a unique identifier number which does not inform the group they are in. The outcome assessor was not aware of which group the participants were allocated in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants had their impacted mandibular third molar (IMTM) extracted according to the standard procedure.
- Experimental Group (Experimental): 20ml of venous blood was collected from each participant in this group into two glass tubes (10ml, A-PRF by Choukroun) and centrifuge to create A-PRF+ using Dou Quattro Choukroun PRF machine with a speed of 1300 rpm in 8 minutes, centrifugal force at the bottom of the tube was RCFmax 208g (RCFmin=113g, RCFav=164g, RCFclot=145g). After the standard extraction procedure, place two A-PRF+ clots in the IMTM socket before suturing.
  Interventions: Combination Product: A-PRF+

INTERVENTIONS:
Combination Product: A-PRF+ — A-PRF+ contributes to accelerating the healing process, more rapid revascularization, and reducing the risk of inflammation at the graft site. It leads to a decrease in the severity of postoperative complications. Many authors have mentioned platelet concentrates as an effective adjunction that improves the healing of hard and soft tissue and decreases pain, swelling, and trismus. However, there are still some controversial results in the literature. Recently, it has been demonstrated that the production of PRF with lower centrifugal force and lower centrifugal time has more potential to release several growth factors and facilitate more favorable healing at the site of the application when compared to standard PRF. Promoting the healing process after tooth extraction using A-PRF+ aims to manage patient discomfort as well as postoperation complications.
  Arms: Experimental Group

SUMMARY:
Objectives: This study aims to evaluate the effects of A-PRF+ on postoperative pain, swelling, and trismus after surgical removal of impacted mandibular third molars.

Method and Materials: A randomized controlled trial with a parallel design was performed on healthy patients with 76 impacted mandibular third molars with similar difficulty level, having needs and indications for extraction. All patients had the same standardized extraction protocol at the Department of Minor Oral Surgery of the National Hospital of Odonto - Stomatology in HCM City. In the study group, patients' blood was collected and centrifugated to produce A-PRF+, then placed in the wisdom tooth sockets after surgery. In the control group, the tooth sockets were curetted and sutured as in standard protocol. Pain value was assessed according to the VAS at 2, 4, and 6-hour time points after patients' lower lips stopped feeling numb, and on the 1st, 3rd, and 7th postoperative day; Swelling was evaluated based on the measurement between facial landmarks; Trismus was assessed based on the distance between incisal edges of upper central incisor and lower incisor during maximum mouth opening on the 3rd and 7th postoperative days. Data obtained were statistically analyzed.

DETAILED DESCRIPTION:
The study was a parallel randomized controlled trial on patients having impacted mandibular third molar (IMTM) extraction. This study was performed at the Department of Minor Oral Surgery in the National Hospital of Odonto - Stomatology in HCM City from October 2019 to April 2021. All patients who had IMTM extraction were examined by the dentists at the Department of Minor Oral Surgery. If IMTM were Montero≥2(7), patients would be referred to the research team. After reviewing the criteria for inclusion and exclusion, the investigators explained to all patients the information about the operation, healing time, and possible complications, and the investigators obtained their informed consent before surgery.

Based on recent research with a power of 80% and α=5%, the investigators calculated the minimum sample size for comparing 2 mean values. The result is each group needs a minimum of 36 participants. The initial sample consisted of 85 in both groups intended to participate in this study at the Department of Minor Oral Surgery in the National Hospital of Odonto - Stomatology in HCM City from October 2019 to April 2021. One patient was excluded from this study because of the ASA PS Index>2. After randomization, one patient in the study group could not collect blood for centrifugation; seven patients were excluded due to lack of compliance (four in the control group, three in the study group). Finally, 76 samples remained in this study (Male 23, Female 53).

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 of age
* Healthy patients (ASA PS index ≤ 2)
* The impacted mandibular third molar (IMTM) had to be in the "deep molars" ≥ 2 (according to Montero classification)
* Absence of acute inflammation and/or infection in the IMTM areas
* No history of NSAID usage four weeks before surgery

Exclusion Criteria:

* Those with systemic conditions or pharmacologic treatments that alter oral microbiota or immunologic response
* Pregnant or breastfeeding women
* Those with the presence of any neoplastic lesion (benign or malignant), clinically or radiologically, at the extraction site or close to the IMTM
* Those with the presence of any radiolucent lesion larger than 1cm at the IMTM
* Those absent of the adjacent teeth
* Lack of compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
VAS index indicating pain value 2 hours immediately after the lips stopped feeling numb | 2 hours immediately after the lips stopped feeling numb
  The pain was evaluated subjectively by suggesting patients mark the severity of pain on the VAS, which ranges from 0 (no pain) to 10 (unbearable pain) in increasing order of pain severity. The patients would record their pain score by marking a point on a straight line; the pain point would be the measured distance from the left end to the point that the patient marked.
VAS index indicating pain value 4 hours immediately after the lips stopped feeling numb | 4 hours immediately after the lips stopped feeling numb
  The pain was evaluated subjectively by suggesting patients mark the severity of pain on the VAS, which ranges from 0 (no pain) to 10 (unbearable pain) in increasing order of pain severity. The patients would record their pain score by marking a point on a straight line; the pain point would be the measured distance from the left end to the point that the patient marked.
VAS index indicating pain value 6 hours immediately after the lips stopped feeling numb | 6 hours immediately after the lips stopped feeling numb
  The pain was evaluated subjectively by suggesting patients mark the severity of pain on the VAS, which ranges from 0 (no pain) to 10 (unbearable pain) in increasing order of pain severity. The patients would record their pain score by marking a point on a straight line; the pain point would be the measured distance from the left end to the point that the patient marked.
VAS index indicating pain value 1 day after surgery | 1 day after surgery
  The pain was evaluated subjectively by suggesting patients mark the severity of pain on the VAS, which ranges from 0 (no pain) to 10 (unbearable pain) in increasing order of pain severity. The patients would record their pain score by marking a point on a straight line; the pain point would be the measured distance from the left end to the point that the patient marked.
VAS index indicating pain value 3 days after surgery | 3 days after surgery
  The pain was evaluated subjectively by suggesting patients mark the severity of pain on the VAS, which ranges from 0 (no pain) to 10 (unbearable pain) in increasing order of pain severity. The patients would record their pain score by marking a point on a straight line; the pain point would be the measured distance from the left end to the point that the patient marked.
VAS index indicating pain value 7 days after surgery | 7 days after surgery
  The pain was evaluated subjectively by suggesting patients mark the severity of pain on the VAS, which ranges from 0 (no pain) to 10 (unbearable pain) in increasing order of pain severity. The patients would record their pain score by marking a point on a straight line; the pain point would be the measured distance from the left end to the point that the patient marked.
Maximum mouth opening at baseline | Before surgery
  The maximum mouth opening (the distance between incisal edges of upper and lower central incisors) difference before and after surgery indicates trismus.
Change in maximum mouth opening between baseline and 3 days after surgery | 3 days after surgery
  The maximum mouth opening (the distance between incisal edges of upper and lower central incisors) difference before and after surgery indicates trismus
Change in maximum mouth opening between baseline and 7 days after surgery | 7 days after surgery
  The maximum mouth opening (the distance between incisal edges of upper and lower central incisors) difference before and after surgery indicates trismus
Mean Facial Landmark Length at baseline | Before surgery
  Preoperatively, patients are marked with landmarks on the face A, B, C, D with an indelible brush to measure facial swelling. A is the canthus of the eye, B is the gonion, C is the tragus, D is the mouth commissure. Patients were seated in a relaxing position with the inferior border of the mandible parallel to the floor. Use a non-elastic ruler that measures preoperative measurements, including AB as vertical swelling score and CD as horizontal swelling score. The patient was re-measured the length size of the two AB and CD that had been marked and measured.
Mean Facial Landmark Length 3 days after operation | 3 days after operation
  Preoperatively, patients are marked with landmarks on the face A, B, C, D with an indelible brush to measure facial swelling. A is the canthus of the eye, B is the gonion, C is the tragus, D is the mouth commissure. Patients were seated in a relaxing position with the inferior border of the mandible parallel to the floor. Use a non-elastic ruler that measures preoperative measurements, including AB as vertical swelling score and CD as horizontal swelling score. The patient was re-measured the length size of the two AB and CD that had been marked and measured.
Mean Facial Landmark Length 7 days after operation | 7 days after operation
  Preoperatively, patients are marked with landmarks on the face A, B, C, D with an indelible brush to measure facial swelling. A is the canthus of the eye, B is the gonion, C is the tragus, D is the mouth commissure. Patients were seated in a relaxing position with the inferior border of the mandible parallel to the floor. Use a non-elastic ruler that measures preoperative measurements, including AB as vertical swelling score and CD as horizontal swelling score. The patient was re-measured the length size of the two AB and CD that had been marked and measured.

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital of Odonto-Stomatology, Ho Chi Minh City, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asutay F, Yolcu U, Gecor O, Acar AH, Ozturk SA, Malkoc S. An evaluation of effects of platelet-rich-fibrin on postoperative morbidities after lower third molar surgery. Niger J Clin Pract. 2017 Dec;20(12):1531-1536. doi: 10.4103/1119-3077.181400. PMID 29378982
- [Background] Gulsen U, Senturk MF. Effect of platelet rich fibrin on edema and pain following third molar surgery: a split mouth control study. BMC Oral Health. 2017 Apr 24;17(1):79. doi: 10.1186/s12903-017-0371-8. PMID 28438151
- [Result] Zhu J, Zhang S, Yuan X, He T, Liu H, Wang J, Xu B. Effect of platelet-rich fibrin on the control of alveolar osteitis, pain, trismus, soft tissue healing, and swelling following mandibular third molar surgery: an updated systematic review and meta-analysis. Int J Oral Maxillofac Surg. 2021 Mar;50(3):398-406. doi: 10.1016/j.ijom.2020.08.014. Epub 2020 Sep 16. PMID 32950350